CLINICAL TRIAL: NCT02396797
Title: Effect Evaluation of a Workplace Intervention Targeting Subjective Health Complaints on Sick Leave, Coping, Health, Job Satisfaction and Social Support
Brief Title: Effect Evaluation of a Workplace Intervention Targeting Subjective Health Complaints
Acronym: atWork
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: The Hospital of Vestfold (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9747
Record Dates: First submitted 2015-02-25; First posted 2015-03-24 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Mental Disorders; Back Pain; Anxiety; Depression
Keywords: Sick leave; Mental Health; Coping; Social Support; Subjective Health Complaints
MeSH Terms: conditions — Mental Disorders; Back Pain; Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The new atWork intervention (Experimental): The intervention group will receive the new atWork intervention, which include a management course and workplace courses for all employees targeting mental health complaints and musculoskeletal complaints.
  Interventions: Behavioral: The new atWork intervention
- The original atWork intervention (Active Comparator): The control group will receive the original atWork intervention, targeting musculoskeletal complaint, and peer support.
  Interventions: Behavioral: The original atWork intervention

INTERVENTIONS:
Behavioral: The new atWork intervention — atWork is a cognitive intervention, and uses a nondirective delivery approach. It does not prescribe any change in lifestyle, but aims at establishing an understanding of common complaints and what to do when pain and health complaints occur. All information is based on the non-injury model, where pain and complaints are not signs of injury caused by wrongdoing or "inappropriate" behavior. The consistent take home message from all parts of the intervention is that keeping up usual activities, including going to work, is beneficial for health and recovery. This group will receive one management course, two workplace courses for all employees targeting mild mental disorders and nonspecific musculoskeletal complaints, and one reflection and review meeting.
  Arms: The new atWork intervention
Behavioral: The original atWork intervention — This group will receive three workplace courses for all employees targeting nonspecific musculoskeletal complaints, and peer support. Peer support involves selecting a peer advisor at the workplace. A peer advisor is a fellow worker without former medical training who as part of the atWork intervention receive more in-depth medical knowledge and training about nonspecific musculoskeletal complaints. The peer advisors role is to give social support and to use their local knowledge of the work place to facilitate staying at work for colleagues with health complaints.
  Arms: The original atWork intervention

SUMMARY:
Mental disorders is one of the most frequent causes of long-term sick leave and disability pensions in Norway, and there is a need for a comprehensive, coordinated response from health and social sectors at the country level to address the burden of mental disorders. The aim of this project is to investigate if a workplace intervention with the aim to increase coping of common mental health complaints and social support can reduce sick leave and improve health.

DETAILED DESCRIPTION:
The atWork intervention was established in 2007 as a new stepped-care approach to musculoskeletal complaints. The intervention consisted of workplace information meetings about musculoskeletal complaint to all employees and peer support. The atWork intervention targeting musculoskeletal complaints reduced sick leave and improved health in a randomized controlled trial. The atWork intervention has now been further developed with the aim to increase effect on sick leave and health. The intervention is now extended to include information about mental health complaints, in addition to a management course. The major societal costs and the negative consequences common mental health complaints induce underline the importance of testing if atWork is an effective way of reducing these consequences.

ELIGIBILITY:
Inclusion Criteria:

* Norwegian primary education unit.
* Participants must be employed in one of the Norwegian primary education units participating in the study.
* Participants must have sufficient Norwegian reading and writing skills.

Exclusion Criteria:

* The organization has received the atWork intervention at an earlier time.
* Participants are not employed in one of the participating organizations.
* Participants do not have sufficient Norwegian reading and writing skills.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1011 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Sick leave, unit level | 1 year
  Sick leave at unit level will be collected through registry data from the Norwegian Labour and Welfare administration (NAV). Thus, we will collect data from all employees in participating units (approximately 100 units), not only the employees responding to questionnaires.

SECONDARY OUTCOMES:
Coping Expectancies; Theoretically Originated Measure of the Cognitive Activation Theory of Stress, TOMCATS | 1 year
  All employees will be asked to complete questionnaires, one before the intervention and at 12 months follow-up.
Health; self-rated health, Subjective Health Complaints Inventory, SHC, Hopkins Symptom Checklist, HSCL-10 | 1 year
Job Satisfaction; Global Job Satisfaction, GJO, Demand-Control-Support-Questionnaire, short Swedish version | 1 year
Social Support; Non directive and Directive Support Survey, NDSS-16. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Torill H Tveito, PhD, Principal Investigator — Uni Research Health
Locations (1):
- Torill Helene Tveito, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnsen TL, Eriksen HR, Baste V, Indahl A, Odeen M, Tveito TH. Effect of Reassuring Information About Musculoskeletal and Mental Health Complaints at the Workplace: A Cluster Randomized Trial of the atWork Intervention. J Occup Rehabil. 2019 Jun;29(2):274-285. doi: 10.1007/s10926-018-9786-6. PMID 29785466
- [Derived] Johnsen TL, Eriksen HR, Indahl A, Tveito TH. Directive and nondirective social support in the workplace - is this social support distinction important for subjective health complaints, job satisfaction, and perception of job demands and job control? Scand J Public Health. 2018 May;46(3):358-367. doi: 10.1177/1403494817726617. Epub 2017 Aug 18. PMID 28820017
- [Derived] Johnsen TL, Indahl A, Baste V, Eriksen HR, Tveito TH. Protocol for the atWork trial: a randomised controlled trial of a workplace intervention targeting subjective health complaints. BMC Public Health. 2016 Aug 19;16(1):844. doi: 10.1186/s12889-016-3515-x. PMID 27542921